CLINICAL TRIAL: NCT06033144
Title: Prevalence of Tapia's Syndrome in Weaning Unit and Associated Factors After Orotracheal Intubation in the ICU
Brief Title: Prevalence of Tapia's Syndrome in Weaning Unit
Acronym: PRESTIO
Status: Recruiting | Type: Observational
Sponsor: Hopital Forcilles (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-A00040-45
Record Dates: First submitted 2023-07-18; First posted 2023-09-13 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Tapia's Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- "Non Tapia group": Patients without Tapia's syndrome
  Interventions: Diagnostic Test: Diagnosis of Tapia's Syndrome
- "Tapia group": Patient with Tapia's syndrome
  Interventions: Diagnostic Test: Diagnosis of Tapia's Syndrome

INTERVENTIONS:
Diagnostic Test: Diagnosis of Tapia's Syndrome — The diagnostic includes :
  * Lingual clinical examination
  * Nasofibroscopy
  * Ultrasonography

SUMMARY:
Tapia syndrome is a rare and poorly understood pathology. It is defined by a concomitant attack of the recurrent (branch of X) and hypoglossal (XII) nerves of peripheral or central origin. It is characterized by the paralysis of a vocal cord and the ipsilateral half of tongue. This damage is most often unilateral but it can also be bilateral. It results in dysphonia and swallowing disorders.

Tapia syndrome is a rare and poorly understood pathology. To date, less than 100 cases have been described in the literature. Previous works are mainly case reports and literature reviews. No prevalence study has been performed to date. Furthermore, disagreements persist regarding the semiology. Indeed, the involvement of the soft palate is not always described.

DETAILED DESCRIPTION:
The main aim of this study was to determine the prevalence of Tapia syndrome in patients admitted to weaning unit after prolonged (>48h) orotracheal intubation in the ICU.

The secondary objectives are to:

* Describe the clinical semiology of Tapia syndrome : lingual involvement, soft palate involvement, impairment of phonation and swallowing ;
* Describe the paraclinical features of Tapia syndrome: recurrent involvement, laryngeal and lingual involvement;
* Identify factors associated with Tapia's syndrome

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized in weaning unit
* Duration of orotracheal intubation in the ICU greater than 48 hours;
* Glasgow score greater than or equal to 13 ;
* Patient at least 18 years of age at the time of inclusion;
* Affiliation with a social security system or beneficiary of such a system ;
* Oral, free, informed and express consent of the patient.

Exclusion Criteria:

* Known history of ENT or neurological pathologies (stroke, head trauma, neurodegenerative disease, brain tumor, ENT cancer);
* Known tumors in the vicinity of the X-nerve pathway;
* Ortner's syndrome (left recurrent nerve compression through the left atrium in mitral stenosis);
* Left lung cancer with subaortic lesion;
* History of cervical adenopathy compressing the X nerve;
* Presence of a cervical or cerebral abscess;
* 24-hour ventilated patient;
* Refusal of the patient or designated trusted person to participate in the study;
* Person subject to a safeguard of justice measure ;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were intubated during more than 48 hours in ICU then tracheostomized and hospitalized in weaning unit.
Sampling Method: Probability Sample
Enrollment: 247 (Estimated)
Dates: Start 2023-04-07 (Actual); Primary Completion 2025-11-07 (Estimated); Study Completion 2027-04-07 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Tapia's syndrome | through study completion, an average of 2 years
  The main objective of this study is to determine the prevalence of Tapia syndrome in patients admitted to the weaning unit after prolonged orotracheal intubation in intensive care. The orotracheal intubation is defined as an intubation longer than 48 hours.

SECONDARY OUTCOMES:
Lingual involvment | through study completion, an average of 2 years
  yes/no/measure of lingual deviation in mm and width of each half of tongue in mm with MEEI software)
Soft palate involvement | through study completion, an average of 2 years
  yes/no
Determining the factors associated with Tapia syndrome | The day of inclusion
  Determining the factors associated with Tapia syndrome : number of prone sessions, duration of intubation (day), duration of mechanical ventilation (day), tracheostomy duration (day), Cormack-Lehane's class, time to tracheostomy cannula removal (day), the time to resume oral feeding (day), number of days in the ICU, number of days in weaning unit, the number of pulmonary infections during the intubation and tracheostomy period, sex, the size of the intubation probe in mm
Dysphonia | After initial swallowing test, maximum 1 week
  GRBAS, maximum time of phonation (s), base frequency (Hz), jitter (%), harmonic noise ratio (dB), vocal range (dB), vocal tessitura (dB)
Dysphagia | through study completion, an average of 2 years
  Functional oral intake scale (Level 1-Nothing by mouth to Level 7-Total oral diet with no restrictions)
Nasofibroscopy | After initial swallowing test, maximum 1 week
  immobility of one or both vocal cords on nasofibroscopy
Ultrasound | After initial swallowing test, maximum 1 week
  hyoid-mandibular distance at rest and during swallowing in cm), tongue thickness at rest in cm, geniohyoidien thickness in mm and area in mm2, echogenicity (Heckmatt score), vallecula stasis (yes/no), stasis in the piriform sinuses (yes/no)

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Forcilles, Férolles-Attilly, Seine-et-Marne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lykoudis EG, Seretis K. Tapia's syndrome: an unexpected but real complication of rhinoplasty: case report and literature review. Aesthetic Plast Surg. 2012 Jun;36(3):557-9. doi: 10.1007/s00266-011-9849-y. Epub 2011 Dec 17. PMID 22179851
- [Background] De Luca P, Cavaliere M, Scarpa A, Savignano L, Cassandro E, Cassandro C, Iemma M. Rehabilitation Protocol for Unilateral Laryngeal and Lingual Paralysis (Tapia Syndrome): Comment About "A Challenging Case of Tapia Syndrome After Total Thyroidectomy" By Ildem Deveci, Mehmet Surmeli, and Reyhan Surmeli. Ear Nose Throat J. 2021 Sep;100(5_suppl):734S-737S. doi: 10.1177/0145561320907433. Epub 2020 Feb 23. PMID 32088986
- [Background] Boga I, Aktas S. Treatment, classification, and review of Tapia syndrome. J Craniofac Surg. 2010 Jan;21(1):278-80. doi: 10.1097/SCS.0b013e3181c678f0. PMID 20098201
- [Background] Caranti A, Bianchini C, Corazzi V, Pelucchi S, Ciorba A. Tapia's Syndrome: keep it in mind! Minerva Anestesiol. 2022 Apr;88(4):293-299. doi: 10.23736/S0375-9393.21.16037-7. PMID 35410105
- [Background] Decavel P, Petit C, Tatu L. Tapia syndrome at the time of the COVID-19 pandemic: Lower cranial neuropathy following prolonged intubation. Neurology. 2020 Aug 18;95(7):312-313. doi: 10.1212/WNL.0000000000010011. Epub 2020 Jun 9. No abstract available. PMID 32518147